CLINICAL TRIAL: NCT04076371
Title: The Treatment Efficacy of Combination Atypical Antipsychotics With Sertraline in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing HuiLongGuan Hospital (Other)
Responsible Party: Principal Investigator, Xiang Yang Zhang, Professor, Beijing HuiLongGuan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CASPsy3
Record Dates: First submitted 2019-07-14; First posted 2019-09-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia
Keywords: schizophrenia; sertraline; olanzapine; risperidone; paliperidone; ziprasidone
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- olanzapine-sertraline combination (Experimental): the patient was prescribed low-dose olanzapine (7.5-10mg/day) combined with low-dose sertraline (50-100mg/day)
  Interventions: Drug: olanzapine-sertraline combination
- only olanzapine (Placebo Comparator): the patient was prescribed moderate to severity dose of olanzapine (12.5-20mg/day)
  Interventions: Drug: only olanzapine
- risperidone-sertraline combination (Experimental): the patient was prescribed low-dose risperidone (2-3.5mg/day) combined with low-dose sertraline (50-100mg/day)
  Interventions: Drug: risperidone-sertraline combination
- only risperidone (Placebo Comparator): the patient was prescribed moderate to severity dose of risperidone (4-6mg/day)
  Interventions: Drug: only risperidone
- paliperidone-sertraline combination (Experimental): the patient was prescribed low-dose paliperidone (3-4.5mg/day) combined with low-dose sertraline (50-100mg/day)
  Interventions: Drug: paliperidone-sertraline combination
- only paliperidone (Placebo Comparator): the patient was prescribed moderate to severity dose of paliperidone (6-9mg/day)
  Interventions: Drug: only paliperidone
- ziprasidone-sertraline combination (Experimental): the patient was prescribed low-dose ziprasidone (60-100mg/day) combined with low-dose sertraline (50-100mg/day)
  Interventions: Drug: ziprasidone-sertraline combination
- only ziprasidone (Placebo Comparator): the patient was prescribed moderate to severity dose of ziprasidone (120-160mg/day)
  Interventions: Drug: only ziprasidone

INTERVENTIONS:
Drug: olanzapine-sertraline combination — the patient was prescribed low-dose olanzapine (7.5-10mg/day) combined with low-dose sertraline (50-100mg/day)
  Other Names: olanzapine-sertraline
  Arms: olanzapine-sertraline combination
Drug: only olanzapine — the patient was prescribed moderate to severity dose of olanzapine (12.5-20mg/day)
  Arms: only olanzapine
Drug: risperidone-sertraline combination — the patient was prescribed low-dose risperidone (2-3.5mg/day) combined with low-dose sertraline (50-100mg/day)
  Other Names: risperidone-sertraline
  Arms: risperidone-sertraline combination
Drug: only risperidone — the patient was prescribed moderate to severity dose of risperidone (4-6mg/day)
  Arms: only risperidone
Drug: paliperidone-sertraline combination — the patient was prescribed low-dose paliperidone (3-4.5mg/day) combined with low-dose sertraline (50-100mg/day)
  Other Names: paliperidone-sertraline
  Arms: paliperidone-sertraline combination
Drug: only paliperidone — the patient was prescribed moderate to severity dose of paliperidone (6-9mg/day)
  Arms: only paliperidone
Drug: ziprasidone-sertraline combination — the patient was prescribed low-dose ziprasidone (60-100mg/day) combined with low-dose sertraline (50-100mg/day)
  Other Names: ziprasidone-sertraline
  Arms: ziprasidone-sertraline combination
Drug: only ziprasidone — the patient was prescribed moderate to severity dose of ziprasidone (120-160mg/day)
  Arms: only ziprasidone

SUMMARY:
A randomized, double-blind trial of the treatment effect of dose-low antipsychotics combined with low-dose sertraline in 1640 schizophrenia patients

DETAILED DESCRIPTION:
OBJECTIVE: This study aimed to evaluate the treatment effect of combination low-dose antipsychotics with low-dose sertraline in 1640 schizophrenia patients

METHODS:

1. atypical antipsychotics and dose: including four atypical antipsychotics to form eight treatment groups: 1) olanzapine (7.5-10mg/day) combined with sertraline (50-100mg/day) group 2) only olanzapine (12.5-20mg/day) group 3) risperidone (2-3.5mg/day) combined with sertraline (50-100mg/day) group 4) only risperidone (4-6mg/day) group 5) paliperidone (3-4.5mg/day) combined with sertraline (50-100mg/day) group 6) only paliperidone (6-9mg/day) group 7) ziprasidone (60-100mg/day) combined with sertraline (50-100mg/day) group 8) only ziprasidone (120-160mg/day) group
2. blood biochemical examination: including blood routine examination, liver function, renal function, thyroid function, glucose and lipid level, prolactin, and related hormones and proteins
3. electrophysiological examination: including electrocardiograph, electroencephalography (EEG), and brain evoked potential
4. scale assessment: each patient was assessed by four clinical psychiatrists using the following scales: 1) psychopathology: positive and negative symptoms scale (PANSS) and clinical global impression scale (CGI-S) 2) emotional symptoms: Hamilton depression rating scale (HAMD) and Hamilton anxiety rating scale (HAMA) 3) social function: personal and social performance scale (PSP) 4) side-effect: treatment emergent side-effect scale (TESS) and rating sale for extrapyramidal side-effect (RESES)
5. blood drug concentration assay: including the drug concentration of olanzapine, risperidone, paliperidone, ziprasidone and sertraline, respectively
6. Weigh gain measurement: to measure height, weight for each patient

The above measurement data were collected at baseline, week4, week8, week 12 and week24.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia by two senior psychiatrists
* Between 18 and 60 years and Han Chinese

Exclusion Criteria:

* A Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV Axis I diagnosis other than schizophrenia
* Documented disease of physical diseases including, but not limited to seizure, epilepsy, aneurysm brain tumor, and stroke, dementia, parkinson's disease, Huntington's disease, multiple sclerosis
* Acute, unstable and/or significant and untreated medical illness (e.g., infection, unstable diabetes, uncontrolled hypertension)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1640 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
changes in psychopathology symptoms on PANSS during antipsychiatric treatment | baseline, week 4, week 8, week 12, and week 24
  The Positive and Negative Syndrome Scale (PANSS) is a well-characterized and widely applied dimensional assessment that reflects a balanced representation of positive and negative syndromes, their differential and general severity of illness. The scales not only measures positive and negative syndromes, but also suggests their differential and general severity of the illness. The items on the PANSS are defined with increasing levels from 1 to 7: 1 = absent, 2 = minimal, 3 = mild, 4 = moderate, 5 = moderate-severe, 6 = severe, and 7 = extreme. Then the PANSS score is totaled by sum up the ratings across different items, the potential range for positive and negative scales are from 7 to 49 whereas the General Psychopathology Scale is ranged between 16 to 112.
changes in depressive symptoms on HAMD during antipsychiatric treatment | baseline, week 4, week 8, week 12, and week 24
  HAMD stands for Hamilton Rating Scale. It is the assessment that designed for examining the treatment significant of depression severity. The general format contains 17 items, 12 of them are scored from 0 to 4 while the rest of them ranges from 0 to 2. The items represented a variety of aspects: Depression mood, Feeling of guilt, Suicide, Insomnia early, Insomnia middle, Insomnia late, Work and activities, Motor retardation, Agitation, Psychic anxiety, Somatic anxiety, Somatic symptoms(gastrointestinal), somatic symptoms(general), Genital symptoms (sexual interest). Hypochondriasis, Weight loss and Insight. So A cut-off score less than or equal to 7 in the HAMD scale defines the symptomatic remission.

SECONDARY OUTCOMES:
changes in electroencephalography examination for brain activity during antipsychiatric treatment | baseline, week 4, week 8, week 12, and week 24
  electroencephalography, or EEG is the physiological method of choice to record the electrical activity generated by the brain via electrodes placed on the scalp surface. For faster application, electrodes are mounted in elastic caps similar to bathing caps, ensuring that the data can be collected from identical scalp positions across all respondents. By analysis of frequency and amplitude of five kind of brain waves(delta, theta, alpha, beta, gamma) , we could detect the synchronized activity of neurons within cortical areas even at sub-second timescales

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoe Lang, Doctor, Study Director — The First Affiliated Hospital of Shanxi Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulholland C, Lynch G, King DJ, Cooper SJ. A double-blind, placebo-controlled trial of sertraline for depressive symptoms in patients with stable, chronic schizophrenia. J Psychopharmacol. 2003 Mar;17(1):107-12. doi: 10.1177/0269881103017001713. PMID 12680747
- [Background] Ros LT. Treatment of postpsychotic depression with sertraline in patients with schizophrenia--own experience. Neuropsychopharmacol Hung. 2006 Oct;8(3):155-6. PMID 17211050
- [Background] Poyurovsky M, Kurs R, Weizman A. Olanzapine-sertraline combination in schizophrenia with obsessive-compulsive disorder. J Clin Psychiatry. 2003 May;64(5):611. doi: 10.4088/jcp.v64n0518c. No abstract available. PMID 12755669
- [Background] Bogers JPAM, Schulte PFJ, Broekman TG, Moleman P, de Haan L. Dose reduction of high-dose first-generation antipsychotics or switch to ziprasidone in long-stay patients with schizophrenia: A 1-year double-blind randomized clinical trial. Eur Neuropsychopharmacol. 2018 Sep;28(9):1024-1034. doi: 10.1016/j.euroneuro.2018.06.005. Epub 2018 Jul 17. PMID 30025751
- [Background] Takekita Y, Koshikawa Y, Fabbri C, Sakai S, Sunada N, Onohara A, Nishida K, Yoshimura M, Kato M, Serretti A, Kinoshita T. Cognitive function and risperidone long-acting injection vs. paliperidone palmitate in schizophrenia: a 6-month, open-label, randomized, pilot trial. BMC Psychiatry. 2016 May 29;16:172. doi: 10.1186/s12888-016-0883-9. PMID 27236412
- [Derived] Guan X, Xiu M, Wu F. Low-dose Olanzapine and Sertraline Combination Therapy for Metabolic Disturbance in Patients with Schizophrenia: A Large-scale, Open-label Randomized Trial. Curr Neuropharmacol. 2025 Nov 3. doi: 10.2174/011570159X395131251008050155. Online ahead of print. PMID 41185506
- [Derived] Lang X, Xue M, Zang X, Wu F, Xiu M, Zhang X. Efficacy of low-dose risperidone in combination with sertraline in first-episode drug-naive patients with schizophrenia: a randomized controlled open-label study. J Transl Med. 2023 Jul 4;21(1):432. doi: 10.1186/s12967-023-04272-7. PMID 37403159
- [Derived] Lang X, Zang X, Yu F, Xiu M. Effects of low-dose combined olanzapine and sertraline on negative and depressive symptoms in treatment-resistant outpatients with acute exacerbated schizophrenia. Front Pharmacol. 2023 Apr 21;14:1166507. doi: 10.3389/fphar.2023.1166507. eCollection 2023. PMID 37153770
- [Derived] Shi H, Xu J, Lang X, Wu HE, Xiu MH, Zhang XY. Comparison of Efficacy and Safety Between Low-Dose Ziprasidone in Combination With Sertraline and Ziprasidone Monotherapy for Treatment-Resistant Patients With Acute Exacerbation Schizophrenia: A Randomized Controlled Trial. Front Pharmacol. 2022 Apr 26;13:863588. doi: 10.3389/fphar.2022.863588. eCollection 2022. PMID 35559243
- [Derived] Zhu C, Guan X, Wang Y, Liu J, Kosten TR, Xiu M, Wu F, Zhang X. Low-Dose Ziprasidone in Combination with Sertraline for First-Episode Drug-Naive Patients with Schizophrenia: a Randomized Controlled Trial. Neurotherapeutics. 2022 Apr;19(3):1037-1046. doi: 10.1007/s13311-022-01242-7. Epub 2022 Apr 25. PMID 35467271
- [Derived] Chen YQ, Li XR, Zhang L, Zhu WB, Wu YQ, Guan XN, Xiu MH, Zhang XY. Therapeutic Response Is Associated With Antipsychotic-Induced Weight Gain in Drug-Naive First-Episode Patients With Schizophrenia: An 8-Week Prospective Study. J Clin Psychiatry. 2021 May 11;82(3):20m13469. doi: 10.4088/JCP.20m13469. PMID 34004092